CLINICAL TRIAL: NCT00624871
Title: Ascorbic Acid Combined With Ibuprofen in Hypoxic Ischemic Encephalopathy: A Randomized Controlled Trial.
Brief Title: Ascorbic Acid and Ibuprofen in Infants With Hypoxic Ischemic Encephalopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Ahmed Helal Elsayed, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2004-MD-thesis-ahmed
Record Dates: First submitted 2008-02-20; First posted 2008-02-28 (Estimated); Last update posted 2008-02-28 (Estimated); Status verified 2008-02

CONDITIONS: Hypoxic Ischemic Encephalopathy; Perinatal Asphyxia
Keywords: Interleukin 1-beta; Interleukin 6; Vitamin C; HIE; neonates
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Ascorbic Acid; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Infants will receive intravenous ascorbic acid and oral ibuprofen for 3 days
  Interventions: Drug: Ascorbic acid (vitamin C); Drug: Ibuprofen
- B (Placebo Comparator): Infants will receive equivalent amount of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ascorbic acid (vitamin C) — IV, 100 mg/kg/day, every day, for 3 days
  Arms: A
Drug: Ibuprofen — PO, 10 mg/kg on day 1, 5 mg/kg/day on days 2 and 3 of life
  Arms: A
Drug: Placebo
  Arms: B

SUMMARY:
Oxygen radicals and inflammation are important causes for brain injury in neonates following perinatal asphyxia. Animal studies demonstrated potential benefits to the brain when using both of vitamin C and ibuprofen. The efficacy of these 2 drugs when combined in protecting the human brain has not been studied. We aimed in this study to test the hypothesis that a combination of anti-oxidants (vitamin C) and anti-inflammatory (ibuprofen) drugs can decrease the brain injury in perinatal asphyxia and improve outcomes when given to infants immediately after birth.

ELIGIBILITY:
Inclusion Criteria:

* Apgar score at 5 minutes < 6
* Profound metabolic or mixed acidosis with pH < 7 in the initial blood gas
* Evidence of encephalopathy such as coma, seizures or hypotonia
* Evidence of multi-system compromise, in addition to encephalopathy

Exclusion Criteria:

* Major congenital anomalies
* Early sepsis
* Gastrointestinal bleeding
* Thrombocytopenia

Max Age: 2 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2004-04; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
DDST-II | 6 months
Neurological Examination | 6 months

SECONDARY OUTCOMES:
Death | On Discharge
Neurological Examination | On Discharge

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elsayed, MD, Principal Investigator — Al-Azhar University; Laila Abd-Rabboh, MD, Study Chair — Al-Azhar University
Locations (1):
- Bab El-Shariya Hospital, Cairo, Cairo Governorate, Egypt